CLINICAL TRIAL: NCT01006356
Title: Cancer Pain Management With Hydromorphone HCl ORal Osmotic System in Korean Cancer Patient: Evaluation of Its Clinical Usefulness in Reduction of Breakthrough Pain Medication Frequency
Brief Title: An Efficacy and Safety Study of Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) in the Reduction of Breakthrough Pain Medication Frequency in Participants With Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015694; 42801PAI4006
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-07

CONDITIONS: Cancer; Pain
Keywords: Hydromorphone hydrochloride Oral Osmotic System; Jurnista
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydromorphone hydrochloride (HCl) oral osmotic system (OROS) (Experimental): Hydromorphone HCl OROS 8 milligram (mg) once daily for 2 weeks.
  Interventions: Drug: Hydromorphone HCl OROS

INTERVENTIONS:
Drug: Hydromorphone HCl OROS — Hydromorphone HCl OROS 8 mg once daily for 2 weeks.

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of hydromorphone hydrochloride (HCl) Oral Osmotic System (OROS) by assessing the extent of reduction of medication frequency for the management of breakthrough pain after the administration of hydromorphone HCl OROS in Korean cancer participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (conducted in more than 1 center), prospective (study following participants forward in time) study. The total duration of study will be 3 weeks. The study consists of 2 periods and 4 visits: screening period (1 week; Visit 1) and treatment period (2 weeks; Visit 2, 3 and 4). During screening period at Visit 1, potential participants will receive previously administered oral opioid analgesic until the second visit and with immediate-release opioid analgesic whenever breakthrough pain is present. During treatment period, from second visit to the fourth visit, participants will receive the hydromorphone HCl OROS once daily for 2 weeks. At Investigator's discretion, participants completing 2 weeks of treatment with study drug could be enrolled into the extension phase of 12-weeks. The dose of study drug is flexible and will be increased or decreased based on the frequency of immediate-release opioid analgesic doses needed to manage pain. At second visit, initial dose of hydromorphone will be determined according to the equivalent analgesic effect conversion tablet (oxycodone 10 milligram [mg] twice daily is equal to hydromorphone HCl 8 mg once daily). The Investigator will increase a participant's daily dose if more than 3 breakthrough pain episodes require rescue medication within a 24 hours period. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Cancer participants administering only strong oral opioid analgesic for cancer pain control
* Participants administering short-acting narcotic analgesics at least twice daily due to breakthrough pain for 3 days just before Visit 2 (Day 1)
* Participants sufficiently capable of complying overall study requirements including participant diary for pain at the discretion of the Investigators
* Abstinent or surgically sterile female participants

Exclusion Criteria:

* Participants with cancer pain who are potentially unresponsive to narcotic analgesics
* Participants with presence or history of drug or alcohol abuse within the past 6 months
* Participants with hypersensitivity to hydromorphone HCl
* Participants with history of colectomy (surgery to remove part or all of the colon)
* Participants with severe digestive tract disease which might interfere with oral analgesic effects, such as dysphagia (trouble swallowing), vomiting, no bowel movement, ileus, and severe enterostenosis that can influence absorption and passing through of oral medication

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydromorphone Hydrochloride Oral Osmotic System: Hydromorphone HCl OROS administered at a dose of 8 milligram once daily for 2 weeks.
Period: Overall Study
Arm/Group | Hydromorphone Hydrochloride Oral Osmotic System
Started | 141
Completed | 99
Not Completed | 42
Not completed — Adverse Event | 6
Not completed — Physician Decision | 1
Not completed — Paticipants did not cooperate | 6
Not completed — Withdrawal by Subject | 1
Not completed — Choice by participants | 2
Not completed — Protocol Violation | 3
Not completed — Other | 23

BASELINE CHARACTERISTICS:
Population: Baseline characteristics was measured for intent-to-treat (ITT) analysis population which was defined as participants who received at least 1 dose of study drug and had available data in the dosing frequency of short-acting narcotic analgesics for treating breakthrough pain at Visit 3 (Day 8).
Groups:
- Hydromorphone HCl OROS: Hydromorphone HCl OROS administered at a dose of 8 milligram once daily for 2 weeks.
Arm/Group | Hydromorphone HCl OROS
Number analyzed (Participants) | 106
Age Continuous [Mean (Standard Deviation); unit: Years] — Age Continuous was measured for intent-to-treat (ITT) analysis population which was defined as participants who received at least 1 dose of study drug and had available data in the dosing frequency of short-acting narcotic analgesics for treating breakthrough pain at Visit 3 (Day 8).
  Years | 57.94 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender was measured for ITT analysis population which was defined as participants who received at least 1 dose of study drug and had available data in the dosing frequency of short-acting narcotic analgesics for treating breakthrough pain at Visit 3 (Day 8).
  Participants
    Female | 37
    Male | 69

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dosing Frequency of Analgesics for Treating Breakthrough Pain
Description: Percentage of participants with decrease in dosing frequency by 33 percent or more in breakthrough pain (acute pain that comes on rapidly despite the use of pain medication) was determined at final visit (Day 15) compared to Baseline (Day 1 - when the administration of study drug was started).
Time Frame: Day 15
Population: The intent-to-treat (ITT) analysis population included all the participants who received at least 1 dose of study drug and had available data in the dosing frequency of short-acting narcotic analgesics for treating breakthrough pain at Day 8. Last observation carried forward (LOCF) was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Hydromorphone HCl OROS
Number analyzed (Participants) | 106
Percentage of Participants | 50.9

2. Secondary Outcome: Frequency of Experiencing Breakthrough Pain
Description: Frequency of experiencing 3 types of breakthrough pain: Idiopathic pain (pain of unknown cause), incidental pain (pain that arises as a result of activity, such as movement of an arthritic joint, stretching a wound) and end-of-dose failure pain was reported.
Time Frame: Day 1 and Day 15
Population: The ITT analysis population included all the as participants who received at least 1 dose of study drug and had available data in the dosing frequency of short-acting narcotic analgesics for treating breakthrough pain at Day 8. LOCF was used.
Measure: Mean (Standard Deviation); unit: Pain episodes per day
Arm/Group | Hydromorphone HCl OROS
Number analyzed (Participants) | 106
Pain episodes per day
  Day 1: Incidental Pain | 1.1 (1.4)
  Day 15: Incidental Pain | 0.8 (1.1)
  Day 1: Idiopathic Pain | 1.8 (1.6)
  Day 15: Idiopathic Pain | 1.2 (1.3)
  Day 1: End-of-dose failure | 1.0 (1.6)
  Day 15: End-of-dose failure | 0.6 (1.0)

3. Secondary Outcome: Change From Baseline in Korean - Brief Pain Inventory (K-BPI) Score at Day 15
Description: K-BPI is an inventory designed to measure the degree of pain severity and the impact of pain in performing daily routines. K-BPI comprises of total 9 items in total, and the ninth item consisting of 7 sub-items is a question asking the degree of disturbance due to pain. The score ranges from 0 to 10, where 0=no pain, 1 to 4=mild pain, 5 to 6=moderate pain and 7 to 10=severe pain.
Time Frame: Baseline and Day 15
Population: The ITT analysis population included all the participants who received at least 1 dose of study drug and had available data in the dosing frequency of short-acting narcotic analgesics for treating breakthrough pain at Day 8. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hydromorphone HCl OROS
Number analyzed (Participants) | 106
Units on a scale
  Baseline | 3.66 (1.29)
  Change at Day 15 | 0.359 (1.191)

4. Secondary Outcome: Pain Intensity Score
Description: Average Pain intensity score experienced by Participant over the last 24 hours of Day 3 and Day 13 was recorded. Pain intensity was measured using numerical rating scale (NRS) ranging from 0=no pain to 10=most severe pain.
Time Frame: Day 3 and Day 13
Population: The ITT analysis population included all the participants who received at least 1 dose of study drug and had available data in the dosing frequency of short-acting narcotic analgesics for treating breakthrough pain at Day 8. LOCF was used. Here 'n' signifies participants evaluable for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hydromorphone HCl OROS
Number analyzed (Participants) | 106
Units on a scale
  Day 3 (8 AM) (n=106) | 3.7 (1.8)
  Day 3 (8 PM) (n=106) | 3.6 (1.8)
  Day 13 (8 AM) (n=103) | 3.3 (1.8)
  Day 13 (8 PM) (n=103) | 3.3 (1.8)

5. Secondary Outcome: Global Assessment of Overall Efficacy of Study Drug by Investigator
Description: Investigator evaluated overall efficacy of study drug and the responses were categorized as: 'ineffective response', 'average response', 'effective response', 'very effectiveresponse', and 'highly effective response'.
Time Frame: Day 15
Population: The ITT analysis population included all the participants who received at least 1 dose of study drug and had available data in the dosing frequency of short-acting narcotic analgesics for treating breakthrough pain at Day 8. LOCF was used. Here "N" signifies participants evaluated for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Hydromorphone HCl OROS
Number analyzed (Participants) | 104
Participants
  Ineffective response | 4
  Average response | 37
  Effective response | 48
  Very effective response | 12
  Highly effective response | 3

6. Secondary Outcome: Global Assessment of Overall Efficacy of Study Drug by Participant
Description: Participants evaluated overall efficacy of study drug and the responses were categorized as: 'ineffective response', 'average response', 'effective response', 'very effectiveresponse', and 'highly effective response'.
Time Frame: Day 15
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Hydromorphone HCl OROS
Number analyzed (Participants) | 104
Participants
  Ineffective | 9
  Average | 31
  Effective | 49
  Very effective | 12
  Highly effective | 3

7. Secondary Outcome: Participant's Preferences Along With Reasons
Description: The number of participants who preferred oral long-acting narcotic analgesics or previously administered oral opioid analgesic were reported along with detailed and specific reasons such as consistent analgesic effect during administration, sleep undisturbed by pain, reduced intake of medication frequency, reduce intake of immediate-release opioid analgesic for breakthrough pain treatment, other and no response, for their preferences. Same participant may have multiple reason for their preference.
Time Frame: Day 15
Population: The ITT analysis population included all participants who received at least 1 dose of study drug and had available data in dosing frequency of short-acting narcotic analgesics for treating breakthrough pain at Day 8. LOCF was used. Here 'N'=participants evaluated for this outcome measure and 'n'=participants who took hydromorphone OROS/oral opioid.
Measure: Number; unit: Participants
Arm/Group | Hydromorphone HCl OROS
Number analyzed (Participants) | 100
Participants
  Hydromorphone OROS:Consistent effect(n=91) | 33
  Oral Opioid: Consistent effect(n=9) | 1
  Hydromorphone OROS: Sleep undisturbed(n=91) | 3
  Hydromorphone OROS:reduced intake frequency(n=91) | 74
  Hydromorphone OROS:reduced intake(n=91) | 29
  Hydromorphone OROS:Other(n=91) | 2
  Oral Opioid: Other(n=9) | 8
  Oral Opioid: No response(n=9) | 1

8. Secondary Outcome: Number of Participants With Clinical Global Impression - Improvement (CGI-I) Score
Description: Investigators evaluated the overall improvement of the participant's condition using CGI scale. The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=greatly improved; 2=somewhat improved; 3=slightly improved; 4=no change; 5=slightly aggravated ; 6=somewhat aggravated; 7=greatly aggarvated.
Time Frame: Day 15
Population: The ITT analysis population included all the participants who received at least 1 dose of study drug and had available data in the dosing frequency of short-acting narcotic analgesics for treating breakthrough pain at Day 8. LOCF was used. Here 'N'=participants evaluated for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Hydromorphone HCl OROS
Number analyzed (Participants) | 104
Participants
  greatly improved | 3
  somewhat improved | 23
  slightly improved | 45
  no change | 30
  slightly aggravated | 1
  somewhat aggravated | 2

9. Secondary Outcome: European Organisation for Research and Treatment of Cancer Quality of Life (EQRTC QLQ-C30) Score
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties) which are based on 4-point scale (1=Not at all to 4=Very much); and global health status and quality of life scale based on 7-point scale (1=very poor to 7=Excellent). All scales and items are averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptomatology or problems.
Time Frame: Day 1 and Day 15
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Hydromorphone HCl OROS
Number analyzed (Participants) | 106
Units on a Scale
  Day 1: Trouble in strenuous activities (n=106) | 3.00 (0.79)
  Day 15: Trouble in strenuous activities (n=106) | 3.07 (0.84)
  Day 1: Trouble in long walk (n=106) | 2.98 (0.78)
  Day 15: Trouble in long walk (n=106) | 3.18 (0.79)
  Day 1: Trouble in short walk outside house (n=106) | 1.98 (0.93)
  Day 15: Trouble in short walk outside house(n=106) | 2.22 (0.99)
  Day 1: Stay in bed/chair (n=106) | 2.64 (0.83)
  Day 15: Stay in bed/chair (n=106) | 2.71 (0.78)
  Day 1: Need help in usual activities (n=106) | 1.56 (0.84)
  Day 15: Need help in usual activities (n=106) | 1.72 (0.95)
  Day 1: Limitation in work/other activites (n=106) | 2.58 (0.81)
  Day 15: Limitation in work/other activites (n=106) | 2.66 (0.84)
  Day 1:Limitation-hobbies/leisure activites(n=106) | 2.56 (0.85)
  Day 15:Limitation-hobbies/leisure activites(n=106) | 2.61 (0.85)
  Day 1: Short of breath (n=106) | 2.02 (0.86)
  Day 15: Short of breath (n=106) | 2.04 (0.87)
  Day 1: Had pain (n=106) | 2.90 (0.74)
  Day 15: Had pain (n=106) | 2.66 (0.79)
  Day 1: Needs rest (n=105) | 2.74 (0.81)
  Day 15: Needs rest (n=105) | 2.78 (0.75)
  Day 1: Trouble in sleeping (n=106) | 2.18 (0.90)
  Day 15: Trouble in sleeping (n=106) | 2.13 (0.87)
  Day 1: Felt weak (n=106) | 2.50 (0.77)
  Day 15: Felt weak (n=106) | 2.52 (0.78)
  Day 1: Apetite loss (n=106) | 2.27 (0.91)
  Day 15: Apetite loss (n=106) | 2.41 (0.94)
  Day 1: Felt nauseated (n=106) | 1.75 (0.83)
  Day 15: Felt nauseated (n=106) | 1.85 (0.90)
  Day 1: Vomitting (n=106) | 1.29 (0.53)
  Day 15: Vomitting (n=106) | 1.24 (0.51)
  Day 1: Constipation (n=106) | 2.15 (0.99)
  Day 15: Constipation (n=106) | 2.08 (0.96)
  Day 1: Diarrhea (n=106) | 1.34 (0.65)
  Day 15: Diarrhea (n=106) | 1.18 (0.47)
  Day 1: Tired (n=106) | 2.62 (0.79)
  Day 15: Tired (n=106) | 2.51 (0.78)
  Day 1:Pain interference - daily activities(n=106) | 2.69 (0.85)
  Day 15:Pain interference - daily activities(n=106) | 2.60 (0.81)
  Day 1: Difficulty in concentrating (n=106) | 2.10 (0.84)
  Day 15: Difficulty in concentrating (n=106) | 2.13 (0.85)
  Day 1: Felt tensed (n=106) | 1.95 (0.76)
  Day 15: Felt tensed (n=106) | 2.01 (0.77)
  Day 1: Worried (n=106) | 2.12 (0.78)
  Day 15: Worried (n=106) | 2.16 (0.81)
  Day 1: Felt irritated (n=106) | 2.22 (0.83)
  Day 15: Felt irritated (n=106) | 2.20 (0.86)
  Day 1: Felt depressed (n=106) | 2.07 (0.82)
  Day 15: Felt depressed (n=106) | 1.94 (0.88)
  Day 1: Difficulty in remembering (n=104) | 2.02 (0.87)
  Day 15: Difficulty in remembering (n=104) | 1.95 (0.84)
  Day 1: Interference in family life (n=106) | 2.47 (0.88)
  Day 15: Interference in family life (n=106) | 2.59 (0.87)
  Day 1: Interference in social life (n=106) | 2.58 (0.88)
  Day 15: Interference in social life (n=106) | 2.60 (0.90)
  Day 1: Economical difficulties (n=106) | 2.58 (0.82)
  Day 15: Economical difficulties (n=106) | 2.51 (0.81)
  Day 1: Global health status (n=106) | 3.42 (1.01)
  Day 15: Global health status (n=106) | 3.42 (1.15)
  Day 1: Quality of life (n=106) | 3.47 (1.04)
  Day 15: Quality of life (n=106) | 3.44 (1.08)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 15
Description: Safety population included 107 participants who administered the study drug more than once and were considered to have data for safety analysis.
Arm/Group | Hydromorphone HCl OROS
Serious Adverse Events (participants affected / at risk) | 33/107
Other Adverse Events (participants affected / at risk) | 95/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Hydromorphone HCl OROS (N=107)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/106
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases tobone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Asthenia (General disorders) | 7
Disease progression (General disorders) | 5
Fatigue (General disorders) | 2
Death (General disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Mallory-weisssyndrome (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Comahepatic (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydromorphone HCl OROS (N=107)
Constipation (Gastrointestinal disorders) | 55 (61)
Nausea (Gastrointestinal disorders) | 34 (36)
Vomiting (Gastrointestinal disorders) | 25 (28)
Diarrhoea (Gastrointestinal disorders) | 12 (13)
Dizziness (Nervous system disorders) | 45 (53)
Asthenia (General disorders) | 43 (45)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (30)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No